CLINICAL TRIAL: NCT03748940
Title: A Study to Investigate the Tolerability of Subcutaneous Injections of LY3074828 Compared to Placebo
Brief Title: Study of LY3074828 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 17097; I9O-MC-AABC (Other: Eli Lilly and Company); 2018-000773-68 (EudraCT Number)
Record Dates: First submitted 2018-09-28; First posted 2018-11-21 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Healthy
MeSH Terms: interventions — mirikizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Part A: Placebo (Placebo Comparator): Placebo administered subcutaneously (SC)
  Interventions: Drug: Placebo
- Part A: LY3074828 (Experimental): LY3074828 administered SC
  Interventions: Drug: LY3074828
- Part B: Placebo (Placebo Comparator): Placebo administered SC
  Interventions: Drug: Placebo
- Part B: LY3074828 (Experimental): LY3074828 administered SC
  Interventions: Drug: LY3074828
- Part B: LY900021 (Experimental): LY900021 (LY3074828 + LY9999QS) administered SC
  Interventions: Drug: LY900021

INTERVENTIONS:
Drug: LY3074828 — Administered SC
  Arms: Part A: LY3074828; Part B: LY3074828
Drug: Placebo — Administered SC
  Arms: Part A: Placebo; Part B: Placebo
Drug: LY900021 — Administered SC
  Arms: Part B: LY900021

SUMMARY:
The purpose of this study is to evaluate different concentrations and formulations of LY3074828 compared to placebo ("dummy drug").

The study will consist of 2 parts: Part A and Part B. Screening is required within 28 days prior to the start of each study part. For each participant in Part A and Part B, the total duration of the clinical trial will be approximately 16 weeks, including screening.

ELIGIBILITY:
Inclusion Criteria:

- Have venous access sufficient to allow for blood sampling and administration of investigational product

Exclusion Criteria:

* Must not have an average weekly alcohol intake that exceeds 28 units per week (males) and 21 units per week (females)
* Must not show evidence of active or latent tuberculosis (TB)
* Must not have received live vaccine(s) (including attenuated live vaccines and those administered intranasally) within 1 month of screening or intend to receive during the study
* Must not be immunocompromised
* Must not have known hypersensitivity to hyaluronidases
* Must not have received treatment with biologic agents (e.g. monoclonal antibodies, including marketed drugs) within 3 months or 5 half-lives (whichever is longer) prior to dosing
* Must not have significant allergies to humanized monoclonal antibodies
* Must not have clinically significant multiple or severe drug allergies, intolerance to topical corticosteroids, or severe post treatment hypersensitivity reactions
* Must not have had lymphoma, leukemia, or any malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years
* Must not have had breast cancer within the past 10 years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2019-06-18 (Actual); Study Completion 2019-06-18 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) Pain Score | Within 1-minute post injection
  The pain VAS is a participant administered single item scale designed to measure pain using a 0-100 millimeter (mm) horizontal VAS. Overall severity of participant's pain is indicated by placing a single mark on the scale from 0 mm (no pain) to 100 mm (severe pain).

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Covance Clinical Research Ltd, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No